CLINICAL TRIAL: NCT02749396
Title: Pregnancy Outcomes in Multiple Sclerosis Populations Exposed and Unexposed to Interferon β - a Register-based Study in the Nordic Countries
Brief Title: EPID Multiple Sclerosis Pregnancy Study
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: EPID Research (Unknown); Biogen (Industry); Merck Serono Europe Ltd (Unknown); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18219
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b; Interferon beta-1a; peginterferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- IFN-β / Cohort 1: Exposure to IFN-β only
  Interventions: Drug: Betaseron (Interferon beta-1b, BAY86-5046), Bayer HealthCare AG; Drug: Extavia (interferon beta-1b), Novartis Pharma AG; Drug: Rebif (interferon beta-1a), Merck Serono Europe Ltd; Drug: Plegridy (peginterferon beta-1a), Biogen Idec Ltd; Drug: Avonex (interferon beta-1a), Biogen Idec Ltd
- IFN-β + other MSDMDs / Cohort 2: Women with MS exposed to IFN-β regardless of exposure to other MSDMDs
  Interventions: Drug: Betaseron (Interferon beta-1b, BAY86-5046), Bayer HealthCare AG; Drug: Extavia (interferon beta-1b), Novartis Pharma AG; Drug: Rebif (interferon beta-1a), Merck Serono Europe Ltd; Drug: Avonex (interferon beta-1a), Biogen Idec Ltd; Drug: MSDMDs other than Betaseron (Interferon beta-1b, BAY86-5046)
- No MSDMDs / Cohort 3: Women with MS exposed with no exposure to any MSDMDs
  Interventions: Other: No MSDMDs therapy (control)
- No IFN-β + other MSDMDs / Cohort 4: Women with MS exposed to IFN-β exposure regardless of exposure to other MSDMDs
  Interventions: Drug: MSDMDs other than Betaseron (Interferon beta-1b, BAY86-5046)
- Other MSDMDs / Cohort 5: Women with MS exposed to other MSDMD only excluding IFN-β or glatiramer acetate (Copaxone) or dimethyl fumarate (Tecfidera)
  Interventions: Drug: MSDMDs other than Betaseron (Interferon beta-1b, BAY86-5046)
- Control / Cohort 6: Women from the general population without MS

INTERVENTIONS:
Drug: Betaseron (Interferon beta-1b, BAY86-5046), Bayer HealthCare AG — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β + other MSDMDs / Cohort 2; IFN-β / Cohort 1
Drug: Extavia (interferon beta-1b), Novartis Pharma AG — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β + other MSDMDs / Cohort 2; IFN-β / Cohort 1
Drug: Rebif (interferon beta-1a), Merck Serono Europe Ltd — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β + other MSDMDs / Cohort 2; IFN-β / Cohort 1
Drug: Plegridy (peginterferon beta-1a), Biogen Idec Ltd — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β / Cohort 1
Drug: Avonex (interferon beta-1a), Biogen Idec Ltd — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β + other MSDMDs / Cohort 2; IFN-β / Cohort 1
Drug: MSDMDs other than Betaseron (Interferon beta-1b, BAY86-5046) — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: IFN-β + other MSDMDs / Cohort 2; No IFN-β + other MSDMDs / Cohort 4; Other MSDMDs / Cohort 5
Other: No MSDMDs therapy (control) — Information will be obtained from the databses DPP (FIN) and MBR (SWE, NOR)
  Groups: No MSDMDs / Cohort 3

SUMMARY:
Multiple Sclerosis (MS) is the most common chronic neurologic disability in young adult females in their childbearing ages. Little evidence is available regarding the association between exposure to IFN-beta (β) products and adverse pregnancy outcomes. Therefore the four marketing holders of IFN-β are conducting a European-wide IFN-β pregnancy registry. Additionally, the Committee for Medicinal Products for Human Use (CHMP) has requested a study to enable identification of pregnancy outcomes in the MS population unexposed to IFN-β products for comparison with the ongoing European IFN-β Pregnancy Registry.

DETAILED DESCRIPTION:
Information will be obtained from the Drugs and Pregnancy Project database (DPP - FIN) and the Medical Birth Register (MBR - SWE, NOR). The Finnish DPP and Norwegian MBR include information on all stillbirths of foetuses with a birth weight of at least 500 g or with a gestational age of at least 22+0 Gestational Week (GW). The Swedish MBR includes data on stillbirths after 28 GW

The estimated number of pregnancies in MS patients needed is 1671, encompassing data from:

i) FIN: 1 January 1996 - 31 December 2014; ii) SWE: 1 July 2005 - 31 December 2014; iii) NOR: 1 January 2004 - 31 December 2014.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had a pregnancy with a recorded outcome consisting of an induced abortion, spontaneous abortion, ectopic pregnancy, or birth during the study period in FIN, SWE or NOR with the event being documented in the relevant databases.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target study population consists of Finnish, Swedish and Norwegian women diagnosed with MS who have been pregnant during the study period from 1996 to 2014. The pregnancy may have resulted in an induced abortion, spontaneous abortion, ectopic pregnancy, stillbirth, or live birth during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2089 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Serious adverse pregnancy outcome due to different regimes of IFN-β exposure defined as a composite endpoint including presence of elective Termination of Pregnancy due to Foetal Anomaly (TOPFA), Major Congenital Anomaly (MCA) or stillbirth | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
Elective TOPFA for other reasons than IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
Elective termination for other reasonsthan IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
Stillbirth due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
Live birth while different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
MCA due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Cohort 1: Exposure to IFN-β only Cohort 2: All patients with IFN-β exposure regardless of exposure to other MS Disease Modifying Drug (MSDMDs) Cohort 3: No exposure to any MSDMDs Cohort 4: All patients with no IFN-β exposure regardless of exposure to other MSDMDs
Comparison of the prevalence of serious adverse pregnancy outcome due to different regimes of IFN-β exposure defined as a composite endpoint including elective TOPFA, MCA or stillbirth | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
Comparison of the prevalence of elective termination for other reasons than due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
Comparison of the prevalence of stillbirth due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
Comparison of the prevalence of live birth due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
Comparison of the prevalence of MCA due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
Comparison of the prevalence of Elective TOPFA due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3) and
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)

SECONDARY OUTCOMES:
Comparison of the prevalence of ectopic pregnancies due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3),
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
  3. Women with MS exposed to IFN-β regardless of exposure to other MSDMDs (cohort 2) vs. unexposed to any MSDMDs (cohort 3)
Comparison of the prevalence of spontaneous abortions due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  1. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to any MSDMDs (cohort 3),
  2. Women with MS exposed to IFN-β only (cohort 1) vs. unexposed to IFN-β regardless of exposure to other MSDMDs (cohort 4)
  3. Women with MS exposed to IFN-β regardless of exposure to other MSDMDs (cohort 2) vs. unexposed to any MSDMDs (cohort 3)
Prevalence of elective TOPFA stratified by specific patient characteristics | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Patient characteristics:
  country, year of pregnancy outcome, chronic diseases, exposure to any teratogenic medications, time since MS diagnosis, duration of MS treatment, maternal age, gestational age, weight of the newborn
Prevalence of stillbirth stratified by specific patient characteristics | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Patient characteristics: country, year of pregnancy outcome, chronic diseases, exposure to any teratogenic medications, time since MS diagnosis, duration of MS treatment, maternal age, gestational age, weight of the newborn
Prevalence of live birth stratified by specific patient characteristics | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Patient characteristics: country, year of pregnancy outcome, chronic diseases, exposure to any teratogenic medications, time since MS diagnosis, duration of MS treatment, maternal age, gestational age, weight of the newborn
Prevalence of MCA stratified by specific patient characteristics | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Patient characteristics: country, year of pregnancy outcome, chronic diseases, exposure to any teratogenic medications, time since MS diagnosis, duration of MS treatment, maternal age, gestational age, weight of the newborn
Comparison of the prevalence of ectopic pregnancies due to different regimes of IFN-β exposure | Retrospective Data analysis: MS patients data encompassing approximately 19 years
  Patient characteristics: country, year of pregnancy outcome, chronic diseases, exposure to any teratogenic medications, time since MS diagnosis, duration of MS treatment, maternal age, gestational age, weight of the newborn

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Finland